CLINICAL TRIAL: NCT03595293
Title: Functional Near Infrared Spectroscopy-based Neurofeedback to Reduce Relapse in Prescription Opioid/Alcohol Use Disorders
Brief Title: fNIRs-based Neurofeedback to Reduce Relapse in pOUD/AUD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 related delays made initiation of the project untenable
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sue Grigson, Professor and Chair, Department of Neural and Behavioral Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8203
Record Dates: First submitted 2018-06-29; First posted 2018-07-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder; Alcoholism; Prescription Drug Dependence; Opioid-use Disorder; Neurofeedback
Keywords: Prescription Opioid Use Disorder; Alcohol Use Disorder; Functional Near-infrared Spectroscopy; Treatment Outcome; Resisting Craving
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental Group for AUD Patients (Experimental): Patients will undergo six NFB sessions from the rDLPFC using a closed-loop fNIRs-based system. During each session, participants will walk through a maze on a computer screen three times. Each maze consists of alternating 30-second rest and 30-second active blocks. During each active block, the participant will come into visual contact with an alcohol image, blocking them from progressing through the maze. When patients encounter the alcohol image and they increase activity in their rDLPFC, the image in the maze will decrease in size and vice versa. The size of the alcohol image can fluctuate throughout each thirty second active block as the raw fNIRs signal from the rDLPFC will be sampled every 500 milliseconds using COBI studio software.
  Interventions: Device: fNIRs-based Neurofeedback
- Sham Feedback Group for AUD Patients (Sham Comparator): Patients will undergo six sham feedback sessions from the skin over the zygomatic arch using a closed-loop fNIRs-based system. During each session, participants will walk through a maze on a computer screen three times. Each maze consists of alternating 30-second rest and 30-second active blocks. During each active block, the participant will come into visual contact with an alcohol image, blocking them from progressing through the maze. When participants encounter the alcohol image and they increase blood supply over the zygomatic area, the image will decrease in size and vice versa. The size of the alcohol image can fluctuate throughout each thirty second active block as the raw fNIRs signal from the zygomatic area will be sampled every 500 milliseconds using COBI studio software.
  Interventions: Device: Sham feedback
- Experimental Group for pOUD Patients (Experimental): Patients will undergo six NFB sessions from the rDLPFC using a closed-loop fNIRs-based system. During each session, participants will walk through a maze on a computer screen three times. Each maze consists of alternating 30-second rest and 30-second active blocks. During each active block, the participant will come into visual contact with a pill image, blocking them from progressing through the maze. When patients encounter the pill image and they increase activity in their rDLPFC, the image in the maze will decrease in size and vice versa. The size of the pill image can fluctuate throughout each thirty second active block as the raw fNIRs signal from the rDLPFC will be sampled every 500 milliseconds using COBI studio software.
  Interventions: Device: fNIRs-based Neurofeedback
- Sham Feedback Group for pOUD Patients (Sham Comparator): Patients will undergo six sham feedback sessions from the skin over the zygomatic arch using a closed-loop fNIRs-based system. During each session, participants will walk through a maze on a computer screen three times. Each maze consists of alternating 30-second rest and 30-second active blocks. During each active block, the participant will come into visual contact with a pill image, blocking them from progressing through the maze. When participants encounter the pill image and they increase blood supply over the zygomatic area, the image will decrease in size and vice versa. The size of the pill image can fluctuate throughout each thirty second active block as the raw fNIRs signal from the zygomatic area will be sampled every 500 milliseconds using COBI studio software.
  Interventions: Device: Sham feedback

INTERVENTIONS:
Device: fNIRs-based Neurofeedback — Patients receive fNIRs-based neurofeedback from the rDLPFC to allow them to modify activation within this area.
  Arms: Experimental Group for AUD Patients; Experimental Group for pOUD Patients
Device: Sham feedback — Patients receive fNIRs-based sham feedback from the left zygomatic area to allow them to modify activation within this area.
  Arms: Sham Feedback Group for AUD Patients; Sham Feedback Group for pOUD Patients

SUMMARY:
This study will examine the impact of functional near-infrared spectroscopy-based neurofeedback to a region within the brain's prefrontal cortex involved with self-regulation of resisting craving in alcohol use and prescription opioid use disorder patients. Participants will be asked to complete two cue reactivity tasks, six sessions of neurofeedback training as well as craving visual analog scales and self-efficacy questionnaires throughout a two-week period of their time in residential treatment at the Caron Treatment Center. They will be followed for 90 days after treatment completion at Caron to assess the impact neurofeedback had on their ability to remain sober once patients are living back in the "real world".

ELIGIBILITY:
Inclusion Criteria:

* sex: male or female
* Age: greater than or equal to 18 years
* Caron Treatment Center residential patients with alcohol use disorder, moderate to severe (equivalent to Alcohol Dependence in DSM-IV-TR), or prescription opioid use disorder (pOUD)
* Fluent in written and spoken English
* Patients who are right-handed
* Valid email address and reliable internet access after leaving the Caron Treatment Center

Exclusion Criteria:

* Patients who are concurrently receiving a psychoactive drug for the treatment of an Axis I disorder.
* Patients with current major depressive disorder or schizophrenia, bipolar disorder, post-traumatic stress disorder, or a history of traumatic brain injury.
* Decisional impairment
* Adults unable to consent
* Women who are pregnant
* Prisoners
* Patients who are left-handed
* No reliable email addresses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Improved capacity to increase neural activity in response to alcohol/pill cues in the rDLPFC measured by the change in the blood-oxygen level dependent (BOLD) signal | First two weeks of protocol
Increase in fNIRs signal response to pill/alcohol cues from pre-to-post neurofeedback sessions. | First two weeks of protocol
  Increase in neural activation in the rDLPFC when viewing alcohol cues from the first neurofeedback session to the sixth (last) session.
Higher levels of abstinence 90-days post-residential treatment completion as assessed by the 7-day timeline followback questionnaires. | First 90 days after treatment completion at Caron Treatment Center
  7-day timeline followback questionnaire will be sent out every week for 12 weeks to assess abstinence

SECONDARY OUTCOMES:
Change in self-reported self-efficacy from pre-to-post neurofeedback sessions assessed via the brief situational confidence questionnaire. | First two weeks of protocol
  Before and after each neurofeedback session, participants will complete a brief situational confidence questionnaire
Change in self-reported craving from pre-to-post neurofeedback sessions assessed via a 100-point craving visual analog scale. | First two weeks of protocol
  Before and after each neurofeedback session, participants will complete a 100-point craving visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S Grigson, PhD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.